CLINICAL TRIAL: NCT02459197
Title: A Proof of Concept Study to Investigate the Effect of T4P1001 Treatment in Patients With Peripheral Neuropathic Pain or Osteoarthritic Pain of Knee or Hip
Brief Title: A Proof of Concept Study to Investigate the Effect of a New Treatment in Patient With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tools4Patient (Other)
Collaborators: International Drug Development Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: T1001-02
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Peripheral Neuropathies; Osteoarthritis
Keywords: Pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- T4P1001 (Active Comparator)
  Interventions: Behavioral: Heat Pain Stimuli A; Behavioral: Positive Video; Drug: Administration of T4P1001 capsules
- Placebo (Sham Comparator)
  Interventions: Behavioral: Heat Pain Stimuli B; Behavioral: Neutral Video; Drug: Administration of Placebo capsules

INTERVENTIONS:
Behavioral: Heat Pain Stimuli A
  Arms: T4P1001
Behavioral: Heat Pain Stimuli B
  Arms: Placebo
Behavioral: Positive Video
  Arms: T4P1001
Behavioral: Neutral Video
  Arms: Placebo
Drug: Administration of T4P1001 capsules — This treatment is given as add-on therapy to patient's regular analgesic treatment
  Arms: T4P1001
Drug: Administration of Placebo capsules — This treatment is given as add-on therapy to patient's regular analgesic treatment
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial conducted in patients suffering from chronic pain is to study the relationship between individual patients' profile and their analgesic response

ELIGIBILITY:
Inclusion Criteria:

* Are men or women of at least 18 years of age
* Diagnosed with Peripheral Neuropathic Pain (PNP) or knee or hip pain attributed to Osteoarthritis (OA) since at least 6 months
* Affiliated with national welfare
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by the relevant Ethics Committee (EC) governing the study sites
* Patients will be required to report pain with a score between 4 and 8 inclusive on the mean Average Pain Score (APS) during the baseline period preceding randomization and to have completed at least 10 days of pain assessments in their diary between Visit 1 and Visit 2. If more than 10 days were completed, the mean APS will be calculated on the last 10 ones.

Inclusion Disease Criteria:

* Diagnosis criterium for PNP: Patient with chronic PNP supported by a distinct neuroanatomical plausible distribution with sensory signs and symptoms, and consecutive to one of the following causes: a traumatic event, a surgical procedure (excluding limb amputation), radiculopathy, post- herpetic or post- zoster neuralgia, diabetic polyneuropathy or post chemotherapy. Diagnosis will have to be confirmed by the DN4 questionnaire at the screening visit (pain is considered as neuropathic if DN4 score ≥ 4)
* Diagnosis criterium for OA: Patient with a unilateral or bilateral OA of the knee or hip diagnosed according to the American College of Rheumatology (ACR) criteria based on clinical and radiographic evidence (Altman et al. 1986). The clinical diagnosis of OA will be confirmed by the ACR clinical and radiographic criteria for classification of idiopathic OA of the knee or hip based upon the following criteria:

  1. Knee or hip pain as an average at least half of the time for the last 3 months before screening visit
  2. At least 1 of the following 3 conditions: Age > 50 or morning stiffness < 30 minutes or crepitus
  3. Kellgren and Lawrence grade > 1 as assessed if possible by an X-ray of the referred joint to confirm the diagnosis. If considered medically required by the Investigator based on patient needs and as part of regular patient management, a new anterior-posterior view X- ray should be obtained and reviewed by Investigator or his delegates to verify that the patient meets the disease diagnostic criteria

Exclusion Criteria:

* Patient changed his/her " regular analgesic therapy " for PNP or OA in the last 4 weeks prior to Visit 1 or during the study.
* Patient's regular analgesic treatment for PNP or OA consists of more than 2 different treatments, with neurostimulation being considered as an analgesic treatment for PNP.
* Patient reported unvariable APS and WPS scores between Visit 1 and Visit 2 (systematically the same APS score and the same WPS score reported).
* Use or plan to use non-topical corticosteroids during the study.
* Have initiated (or plan to initiate) a program (or modify an existing program in frequency and/or intensity) of physiotherapy or behavioral therapy such as pain self-management, hypnosis, sophrology, meditation program within 2 weeks prior to Visit 1 or during the study.
* Pregnant, breastfeeding, or willing to be pregnant within 3 months.
* Patients with a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the patient's participation in the study.
* Uncontrolled epilepsy.
* Any current primary psychiatric condition, including depression or personality disorders (such as Axe II of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV); personality disorders and mental retardation).
* Alcohol dependence or regular use of known drugs of abuse (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, and phencyclidine).
* Any other relevant medical disorder/acute disease state judged by the Investigator as likely to interfere with the trial or represent a risk for the patient.
* Any close relationship with the Investigators or the Sponsor (i.e. belonging to immediate family or subordination link).
* Patient under legal protection, according to the national law.
* Are persons who have previously received T4P1001, have completed or withdrawn from this study or any other study investigating T4P1001.
* Patient currently enrolled in a clinical trial involving use of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study, or in an exclusion period according to the national law.

Exclusion Disease Criteria for PNP patients:

* Neuropathic pain due to trigeminal neuralgia, central pain or phantom limb pain.
* Have initiated, are planning to initiate an electrical stimulation (or neurostimulation) therapy or modify an existing neurostimulation within 4 weeks prior to Visit 1 or during study period.

Exclusion disease criteria for OA patients:

* Non-ambulatory due to OA.
* Use of lower extremity assistive devices other than a cane such as crutches or walker or a knee brace or a "shoe lift" in relation to OA.
* Have used in relation to OA systemic corticosteroids 4 weeks prior to Visit 1; Intra-muscular corticosteroid injections or Intra-articular injection of steroids into the referred knee/hip within 3 months before Visit 1, Intra-articular injection of corticosteroids into any other sites than the referred knee/hip within 4 weeks prior to Visit 1(corticosteroids in topical use are allowed).
* Have used viscosupplementation or intra articular injection of hyaluronic acid in the referred joint within 3 months prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pereira, Study Director — Tools4Patient
Locations (6):
- ATC sa, Liège, Belgium
- France (5):
  - CIC Clermont-Ferrand, CHU Clermont-Ferrand, Clermont-Ferrand
  - Eurofins Optimed, Gières
  - Clinique Breteche, Nantes
  - Institut Curie, Paris
  - Centre d'Evaluation et Traitement de la Douleur, CHU Saint-Etienne, Saint-Etienne

RESULTS

PARTICIPANT FLOW:
Groups:
- T4P1001: Heat Pain Stimuli A
  Positive Video
  Administration of T4P1001 capsules: This treatment is given as add-on therapy to patient's regular analgesic treatment
- Placebo: Heat Pain Stimuli B
  Neutral Video
  Administration of Placebo capsules: This treatment is given as add-on therapy to patient's regular analgesic treatment
Period: Overall Study
Arm/Group | T4P1001 | Placebo
Started | 58 | 56
Completed | 58 | 55
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: 3 patients who completed the study were excluded from the Baseline Analysis Population due to protocol violations. Therefore only 110 patients were included in the Baseline Analysis Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | T4P1001 | Placebo | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.2) | 62.4 (12.1) | 61.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 38 | 65
  Male | 30 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Patient's Change From Baseline of Pain Severity as Measured by the Weekly Means of the Daily Average Pain Scores (APS) During 4 Weeks of Treatment
Description: 11-point Numeric Rating Scale (NRS); the 11 NRS scale ranges from 0 (No pain) to 10 (pain as bad as you can imagine); the baseline APS (weekly mean of the daily average pain score) was computed on the 7 last days before Visit 2 with available APS values; similarly, the end-of-treatment APS (or APS Week 4) was computed on the 7 last days before Visit 4 with available APS values.
Time Frame: Time zero equals baseline (Day-28 to Day-14) up to Day 36
Population: 3 patients who completed the study were excluded from the Analysis Population due to protocol violations. Therefore only 110 patients were included in the Analysis Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 57 | 53
score on a scale | 0.54 (1.92) | 0.95 (1.86)

2. Secondary Outcome: Patient's Change From Baseline of Pain Severity as Measured by the Brief Pain Inventory (BPI)
Description: BPI is a self-reported scale that measures the severity of pain and the interference of pain on function (Charles S. Cleeland © 2009). In the short form of BPI, there are 4 questions assessing worst pain, least pain, actual pain and average pain in the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as bad as you can imagine). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. The interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Time zero equals baseline (Day-28 to Day-14) up to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 56 | 53
score on a scale
  Pain | 0.98 (1.63) | 1.61 (1.49)
  Interference of pain | 1.09 (1.93) | 1.94 (1.71)

3. Secondary Outcome: Patient's Change From Baseline of Investigator and Patient Global Assessment of Changes (IGAC and PGAC)
Description: IGAC and PGAC are subjective evaluations using a NRS with 0 meaning "best condition" and 10 "worst condition"
Time Frame: Time zero equals baseline (Day-28 to Day-14) up to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 57 | 53
score on a scale
  PGAC | 1.11 (2.25) | 2.04 (1.93)
  IGAC | 0.96 (1.82) | 1.83 (1.9)

4. Secondary Outcome: Patient's Change From Baseline of Heat Pain Threshold From Baseline to End of Treatment
Description: celcius degree, arithmetic average of 6 tests.
Time Frame: Time zero equals baseline (Day 1) up to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 57 | 53
°C | -0.05 (3) | -0.67 (3.26)

5. Secondary Outcome: For Osteoarthritic Patients Only: Patient's Change From Baseline of Osteoarthritic Physical Function, Pain and Stiffness as Assessed by Western Ontario and MacMaster (WOMAC) Scales From Baseline to End of Treatment
Description: The WOMAC (Bellamy et al., 1988) is a patient-rated instrument that measures OA symptoms.
  The questionnaire contains 5 pain questions, 2 stiffness questions, and 17 physical function questions (24 questions total). Each question utilizes a 5-points Numeric Rating Scale (NRS) between 0-4; from 0=none to 4=extreme. Range of possible subscale scores: pain=0-20, stiffness=0-8 and physical function=0-68; higher scores for each subscale indicate worse outcomes.
  The WOMAC was completed at each Visit except for Visit 5 by OA patients only.
Time Frame: Time zero equals baseline (Day-28 to Day-14) up to Day 29
Population: Only OA sub-population of patients were included in the Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 28 | 24
score on a scale
  Pain | 2.32 (3.62) | 4.08 (3.13)
  Stiffness | 0.93 (1.59) | 1.67 (1.43)
  Physical function | 6.71 (9.37) | 13.67 (11.53)

ADVERSE EVENTS:
Description: All safety analyses included the 58 PNP patients and the 56 OA patients enrolled into the study. Of note, the PNP patient N-043 and the OA patients O-040 and O-061 completed the study and took the treatment for the entire treatment period but were identified as protocol violators due to inclusion criteria not met.
Arm/Group | T4P1001 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/58 | 1/56
Other Adverse Events (participants affected / at risk) | 14/58 | 13/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T4P1001 (N=58) | Placebo (N=56)
Affect lability (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T4P1001 (N=58) | Placebo (N=56)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3
Headache (Nervous system disorders) | 7 | 7
Somnolence (Nervous system disorders) | 3 | 1
Fatigue (General disorders) | 3 | 5
Nausea (General disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less